CLINICAL TRIAL: NCT01845935
Title: Cryoablation of Venous Vascular Malformations Located in Soft Tissues
Brief Title: Cryoablation of Venous Vascular Malformations
Acronym: CRYOMAV
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHUBX 2012/15
Record Dates: First submitted 2013-04-23; First posted 2013-05-03 (Estimated); Last update posted 2016-08-22 (Estimated); Status verified 2016-08

CONDITIONS: Venous Vascular Malformation
Keywords: Cryoablation; Venous vascular malformation; MRI; safety; pain
MeSH Terms: conditions — Pain | interventions — Needles

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- only one treatment group (Experimental): Patients presenting inoperable venous vascular malformations in soft tissues with indication of cryoablation.
  Interventions: Device: Percutaneous Image-guided Cryoablation (FPRPR3508 IceRod® PLUS Needles)

INTERVENTIONS:
Device: Percutaneous Image-guided Cryoablation (FPRPR3508 IceRod® PLUS Needles) — Treatment consists of a percutaneous cryoablation performed under anesthesia and imaging control.

SUMMARY:
To now, two alternatives for the management of venous vascular malformations are recognized, appropriate to the location, size and patients: sclerosis and surgery. However, sclerosis is effective on symptoms in 80% of cases and excision removes the malformation completely or partially, but it is aggressive and recurrences are common.

DETAILED DESCRIPTION:
In order to propose an additional alternative option, cryoablation has been recently tested with promising results. Therefore, the purpose of this study is to evaluate the safety and efficacy of cryotherapy on venous vascular malformations.

Fourteen patients will be included after discussion in multidisciplinary meeting. Patients will be follow until 6 months to evaluate the safety and the 6 months efficacy on symptoms. A MRI will be perform at 6 months to evaluate the size of ablated zone following RECIST criteria.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years,
* Initial radiological diagnosis of venous or glomovenous vascular malformation proved by Doppler ultrasound and MRI,
* Recurrence of symptoms after initial treatment,
* Symptomatic deformation :pain, tangible mass,functional discomfort
* Recurrence after treatment by surgery or sclerosis
* Cryotherapy considered technically feasible after discussion in multidisciplinary committee,
* Localization at distance from the skin and major neurovascular structures,
* Absence of contra-indication of anaesthesia,
* Signed informed consent,
* Coverage by French social security

Exclusion Criteria:

* Localization of the lesion does not allow the implementation of cryotherapy in adequate conditions: ablation zone too close to the major anatomic structures (nerve),
* TP <50% TCA> 1.5 x control, anticoagulation
* Platelets <90000/mm3,
* Progressive infection
* Patient included in another clinical study,
* Unable to undergo medical tests for geographical, social or psychological,
* Adult under a legal guardianship or unable to consent,
* Pregnancy and breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2013-04; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety of cryoablation by measuring the immediate complications using NCI-CTCAE toxicity scale. | 7 days after cryoablation
To evaluate the safety of cryoablation by measuring the delayed complications using NCI-CTCAE toxicity scale. | 1 month after cryoablation
To evaluate the safety of cryoablation by measuring the delayed complications using NCI-CTCAE toxicity scale. | 2 months after cryoablation
To evaluate the safety of cryoablation by measuring the late complications using NCI-CTCAE toxicity scale. | 6 months after cryoablation

SECONDARY OUTCOMES:
All adverse events using NCI-CTCAE | 7 days, 1 month ,2 months + 6 months after cryoablation
Clinical response (decrease of pain and/or functional discomfort) | 6 months after cryoablation
Imaging response (RECIST 1.1) | 6 months after cryoablation
Quality of life using QLQ-C30 | 2 months & 6 months after cryoablation
Pain using visual analogue scale | 7 days, 1 month ,2 months & 6 months after cryoablation

CONTACTS AND LOCATIONS:
Overall Officials: François Cornelis, MD, Principal Investigator — University Hospital Bordeaux, France; Adelaide Doussau, MD, Study Chair — University Hospital Bordeaux, France
Locations (1):
- University Hospital Bordeaux, France, Bordeaux, France

REFERENCES:
- [Background] Cornelis F, Neuville A, Labreze C, Kind M, Bui B, Midy D, Palussiere J, Grenier N. Percutaneous cryotherapy of vascular malformation: initial experience. Cardiovasc Intervent Radiol. 2013 Jun;36(3):853-6. doi: 10.1007/s00270-012-0434-9. Epub 2012 Jun 22. PMID 22722720
- [Background] Cornelis F, Havez M, Lippa N, Al-Ammari S, Verdier D, Carteret T, Amoretti N, Gangi A, Palussiere J, Hauger O, Grenier N. Radiologically guided percutaneous cryotherapy for soft tissue tumours: A promising treatment. Diagn Interv Imaging. 2013 Apr;94(4):364-70. doi: 10.1016/j.diii.2013.02.001. Epub 2013 Mar 11. PMID 23491212
- [Background] Barza M, Pavan PR, Doft BH, Wisniewski SR, Wilson LA, Han DP, Kelsey SF. Evaluation of microbiological diagnostic techniques in postoperative endophthalmitis in the Endophthalmitis Vitrectomy Study. Arch Ophthalmol. 1997 Sep;115(9):1142-50. doi: 10.1001/archopht.1997.01100160312008. PMID 9298055